CLINICAL TRIAL: NCT05579925
Title: A Multicenter, Single-arm, Open-label Study to Evaluate the Safety, Pharmacokinetics, and Pharmacokinetics of CM310 in Adolescent Subjects With Moderate-to-severe Atopic Dermatitis
Brief Title: A Study of CM310 in Children Patients With Moderate-to-severe Atopic Dermatis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Keymed Biosciences Co.Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CM310-101108
Record Dates: First submitted 2022-10-11; First posted 2022-10-14 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2023-06

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CM310 (Experimental): 600 mg + 300 mg, subcutaneous injection, once every two weeks
  Interventions: Biological: CM310

INTERVENTIONS:
Biological: CM310 — CM310 600 mg + 300 mg, subcutaneous injection

SUMMARY:
This is a multi-center, single arm, open-label study to evaluate safety and primary efficacy in children patients with moderate-to severe atopic dermatis.

ELIGIBILITY:
Inclusion Criteria:

* 12 years ≤ age ≤ 18 years
* With atopic dermatis
* Voluntarily sign the informed consent form

Exclusion Criteria:

* Weight < 30 kg
* Major surgery planed during the study

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 24 (Actual)
Dates: Start 2022-10-07 (Actual); Primary Completion 2023-07-28 (Actual); Study Completion 2023-07-28 (Actual)

PRIMARY OUTCOMES:
Adverse events | at week 14
  Incidence of adverse events.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Children's Hospital Capital Medical University, Beijing, China